CLINICAL TRIAL: NCT06904469
Title: Ostrobothnia Digital Clinic Experiment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Aalto University (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Lauri Sääksvuori, Principal investigator, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: THL/5935/6.02.01/2024
Record Dates: First submitted 2025-03-18; First posted 2025-04-01 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-03

CONDITIONS: Primary Care Provider
Keywords: digital healthcare; telemedicine; digital clinic; primary care; healthcare utilization; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trials, households as clusters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Access to a digital clinic (Experimental): Access to a digital clinic, which offers assessments, diagnoses, follow-up care recommendations, and prescriptions
  Interventions: Other: Access to a digital clinic
- No access to a digital clinic (treatment as usual) (No Intervention): Health care as usual without access rights to a digital clinic

INTERVENTIONS:
Other: Access to a digital clinic — This intervention grants access to a digital clinic that provides chat-based primary care consultations via phone application and website.
  Arms: Access to a digital clinic

SUMMARY:
This randomized controlled trial (RCT) examines the impacts of a publicly provided digital clinic that offers digital primary care services to consumers. This intervention grants access to a public digital clinic that provides chat-based primary care consultations via a mobile phone application and website, including care needs assessment, diagnoses, follow-up care recommendations, and prescriptions. The digital clinic supplements traditional public primary care services, including in-person visits and phone consultations. The trial takes place in Ostrobothnia, Finland, a healthcare district serving a population of 178,000 residents. The investigators will randomize access to the digital clinic at the household level, providing access to 50% of the households. By doing so, the investigators aim to evaluate whether digital services can substitute for, complement, or increase the utilization of traditional primary care, particularly in-person visits or calls to traditional clinics. At the end of the nine-month trial, access to the digital clinic will be expanded to the entire population.

ELIGIBILITY:
Inclusion Criteria for the intervention:

* All residents alive and residing in the region of Ostrobothnia (Finland) on March 14, 2015, AND permanent address observed in the Finnish Population Information System

Exclusion Criteria for the intervention:

* Resides in the city of Kristiinankaupunki OR resides in a household defined as institutionalized care

Exclusion Criteria for the analysis sample:

* The inclusion and exclusion criteria mentioned above AND:
* If an individual from the target population, extracted from the Population Information System, is not observed in Statistics Finland datasets, which is defined as not having a municipality of residence (missing data) at the end of 2024, the investigators will not use that individual in the study population in the analyses because the data do not include have covariates for the individual.
* Age 71 and above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170306 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
The number of in-person visits in public primary care (Y1.1) | From the digital clinic launch to the end of treatment at 9 months
  This outcome includes in-person visits to nurses and physicians in traditional public primary care clinics.

SECONDARY OUTCOMES:
The number of other contacts with traditional public primary care (Y1.2) | From the digital clinic launch to the end of treatment at 9 months
  This outcome includes care needs assessments, remote appointments to nurses and physicians, and professional-to-professional interactions between nurses and physicians in traditional public primary care clinics.
The number of public digital clinic contacts (D.1). | From the digital clinic launch to the end of treatment at 9 months
  This outcome includes care needs assessments, remote appointments to nurses and physicians (via chat and video), and professional-to-professional interactions between nurses and physicians in digital public primary care clinics.

OTHER OUTCOMES:
The total number of public primary care contacts (Y1.3) | From the digital clinic launch to the end of treatment at 9 months
  This outcome includes in-person visits to nurses and physicians, care needs assessments, remote appointments to nurses and physicians, and professional-to-professional interactions between nurses and physicians in digital and traditional public primary care clinics.
Presence or absence of public digital clinic contacts during the follow-up (yes/no) (D.2). | From the digital clinic launch to the end of treatment at 9 months
  This outcome includes care needs assessments, remote appointments to nurses and physicians (via chat and video), and professional-to-professional interactions between nurses and physicians in digital public primary care clinics.
  This outcome is 1 if the person has at least one contact with the public digital clinic during follow-up and 0 if the person has no contact during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mika T Kortelainen, PhD, Study Director — University of Turku and Finnish Institute for Health and Welfare
Locations (1):
- Wellbeing Services County of Ostrobothnia, Vaasa, Finland

IPD SHARING:
Plan to Share IPD: No
The dataset containing individual-level health data and demographic data is regulated under the Act on the Secondary Use of Health and Social Data (552/2019) and cannot be made readily available for the purpose of direct replication. However, access to the data can be obtained by sending requests to the Finnish Social and Health Data Permit Authority, Findata, and to Statistics Finland. The investigators commit to publishing all statistical code and other details of the computations that are sufficient to permit the validation of empirical work. The investigators commit to storing the treatment assignment code and data for future use, allowing interested researchers to construct the full dataset required for further research utilizing the original treatment assignment.

REFERENCES:
- See also: Replication codes (GitHub) — https://github.com/tapiohaa/SoteDataLab/tree/main/ostrobothnia_digital_clinic_experiment
- See also: Pre-analysis plan as of March 28, 2025 — https://osf.io/qepn3